CLINICAL TRIAL: NCT03902730
Title: Lower Limb Muscle Activity and Recruitment Patterns Measured Via Electromyography in Back Squat Variations
Brief Title: Leg Muscle Activity Measured Via Electromyography in Back Squat Variations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mary Hardin-Baylor (Other)
Responsible Party: Principal Investigator, Lemuel W. Taylor IV, Director of Research in HPL, University of Mary Hardin-Baylor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: EMG-1
Record Dates: First submitted 2019-03-26; First posted 2019-04-04 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Surface Electromyography; Muscular Fatigue
Keywords: Electromyography; Resistance trained

STUDY DESIGN:
Intervention Model Description: Participants will complete all four trials in a crossover design. A one week washout period is required between treatments.
Who Masked: Participant
Masking Description: Investigators will randomize treatments for all participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Back Squat Variation One (Other): In a randomized order, traditional back squat will be completed.
  Interventions: Other: Traditional Back Squat
- Back Squat Variation Two (Other): In a randomized order, barefoot back squat will be completed.
  Interventions: Other: Barefoot Back Squat
- Back Squat Variation Three (Other): In a randomized order, box squat will be completed.
  Interventions: Other: Box Squat
- Back Squat Variation Four (Other): In a randomized order, traditional back squat with chains will be completed.
  Interventions: Other: Traditional Back Squat with Chains

INTERVENTIONS:
Other: Traditional Back Squat — Participants will complete traditional back squat in this four treatment crossover design.
  Arms: Back Squat Variation One
Other: Barefoot Back Squat — Participants will complete barefoot back squat in this four treatment crossover design.
  Arms: Back Squat Variation Two
Other: Box Squat — Participants will complete box squat in this four treatment crossover design.
  Arms: Back Squat Variation Three
Other: Traditional Back Squat with Chains — Participants will complete traditional back squat with chains in this four treatment crossover design.
  Arms: Back Squat Variation Four

SUMMARY:
The purpose of the study is to see how different forms of the squat exercise change my body's leg muscle activity. Four forms of the traditional back squat will be used: traditional back squat, barefoot squat, box squat, and traditional back squat with chains.

DETAILED DESCRIPTION:
Resistance exercise has various benefits that promote health and reduce the chance of chronic disease, but the biggest benefit may be found in the effects on maintaining muscle mass throughout the aging process. The implications resistance training has on an individual's ability to function throughout the day with less fatigue whilst performing tasks at an easier level can all be related to improved strength and endurance that comes with resistance training. Furthermore, how the nervous system adapts and sends signals to the working muscles are of great interest as neuromuscular adaptations help in coordination, balance, and agility. Variations of the same style of exercise have been theorized to improve and/or change the adaptations that can occur. Thus, the purpose of this study would be to assess surface electromyography (sEMG) activations on 4 anatomical sites simultaneously during the squat exercise under varying conditions.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be males and females between the ages of 18 - 30 years
* Participant has provided written and dated informed consent to participate
* Participant is willing and able to comply with the protocol
* Participant is apparently healthy and free from disease, as determined by a health history questionnaire
* Participant agrees to abstain from lower body exercise 3 days prior to each testing visit
* Participant has completed at least 1 lower body workout every week for the past 6 months

Exclusion Criteria:

* Participant reports any unusual adverse events associated with this study that in consultation with their physician recommends removal from the study
* Participant begins consumption of new supplement during the timeline of this study
* Participant is unable to refrain from consuming pre-workout supplement prior to testing sessions
* Participant is unwilling to refrain from lower body exercise at least 3 days prior to each testing session

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-09-25 (Actual); Study Completion 2021-09-25 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Mean Peak Muscle Activity Between Four Back Squat Variations | Up to 4 weeks
  Participants will complete 5 sets of 10 repetitions at 70% of their 1 repetition maximum with 1-minute rest in between each set under different variations of the back squat. Each week, participants will be randomly assigned to complete a variation of back squat. Under each variation, surface electromyography recordings will consist of mean peak muscle activity as measured via BIOPAC BSL for the first and last sets of the training protocol. Thus, changes between first and last sets of the training protocol will be assessed for changes as well as comparisons between each variation of back squat to assess changes.

SECONDARY OUTCOMES:
Change from Baseline Mean Muscle Activity Between Four Back Squat Variations | Up to 4 weeks
  Participants will complete 5 sets of 10 repetitions at 70% of their 1 repetition maximum with 1-minute rest in between each set under different variations of the back squat. Each week, participants will be randomly assigned to complete a variation of back squat. Under each variation, surface electromyography recordings will consist of mean muscle activity as measured via BIOPAC BSL for the first and last sets of the training protocol. Thus, changes between first and last sets of the training protocol will be assessed for changes as well as comparisons between each variation of back squat to assess changes.

CONTACTS AND LOCATIONS:
Overall Officials: Lemuel W Taylor IV, PhD, Principal Investigator — UMHB Human Performance Lab
Locations (1):
- UMHB Human Performance Lab, Belton, Texas, United States

IPD SHARING:
Plan to Share IPD: No